CLINICAL TRIAL: NCT04231552
Title: Preoperative Short Course Radiotherapy With Consolidation Chemotherapies and Camrelizumab Followed by Delayed Surgery in Locally Advanced Rectal Cancer
Brief Title: Preoperative Short Course Radiotherapy With Chemotherapy and Camerelizumab in Locally Advanced Rectal Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Chief of gastrointestinal oncology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WUGO-001
Record Dates: First submitted 2020-01-04; First posted 2020-01-18 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer; Radiotherapy; Immunotherapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — camrelizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chemotherapy and PD1 inhibitor (Experimental): CAPOX (2 cycles): Oxaliplatin(130mg/m2) on day 1 of each cylce and Capecitabine:Dose of 2000mg/m2,14days, q3w Camrelizumab (2 cycles): 200mg on day 1 of each cycle, q3w Surgical therapy: the resection (LAR), intersphincteric resection (ISR), or abdominoperineal resection (APR).
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Radiotherapy with CAPOX+ Camrelizumab following surgical therapy Radiation: 25 Gy/5 fractions CAPOX (2 cycles): Oxaliplatin(130mg/m2) on day 1 of each cylce and Capecitabine:Dose of 2000mg/m2,14days, q3w Camrelizumab (2 cycles): 200mg on day 1 of each cycle, q3w Surgical therapy: the resection (LAR), intersphincteric resection (ISR), or abdominoperineal resection (APR)
  Other Names: Radiotherapy with CAPOX+ Camrelizumab following surgical therapy

SUMMARY:
This is a open-label, single-arm study to investigate the safety and efficacy of consolidative chemotherapy with camrelizumab, an anti-PD-1 antibody drug following short course radiotherapy and subsequent surgical therapy in patients with locally advanced resectable rectal cancer.

DETAILED DESCRIPTION:
Patients with locally advanced rectal cancer (cT3-4 or N+) are assigned to receive preoperative 5 × 5 Gy irradiation over 5 days with consolidation chemotherapy consisting two cycles of CAPOX chemotherapy and camrelizumab, an anti-PD-1 antibody drug for two cycles. Subsequent surgical therapy is performed to evaluate the safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who personally provided written consent for participation in the study
2. Treatment-naive patients with rectal cancer, in whom the inferior margin of the tumor is at a distance of 10 cm or less from the AV before CRT
3. Primary rectal cancer histopathologically confirmed to be adenocarcinoma
4. Clinical stage of T3/T4 or N positive and M0,before CRT
5. Patients with the ECOG performance status of 0 or 1 at the time of enrollment
6. Women of childbearing potential who consent to practicing contraception during the period from giving informed consent to at least 23 weeks after the last dose of therapy
7. Male patients who consent to practicing contraception during the period from giving informed consent to at least 31 weeks after the last dose of the study drug

Exclusion Criteria:

1. Patients with recurrent rectal cancer or a history of pelvic radiation
2. Patients with a history of inflammatory bowel disease
3. Patients with a history of pneumonitis or interstitial lung disease
4. Patients with concurrent autoimmune disease or a history of chronic or recurrent autoimmune disease
5. Patients requiring treatment with systemic corticosteroids or immunosuppressants or who have received these treatments within 14 days before enrollment in the study
6. Patients with a history of thyroid dysfunction
7. Patients with a history or finding of cardiovascular risk
8. Patients who are positive for any of the following: HIV1 antibody, HIV2 antibody, HTLV1 antibody
9. Patients who are pregnant or lactating or who may be pregnant
10. Patients with significant unstable mental diseases or other medical diseases that may interfere with the safety of the subjects, obtaining informed consent, or compliance with the procedures for the clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response | 1 year
  Pathological complete response will be evaluated with American Joint Committee on Cancer (AJCC) Cancer Staging

SECONDARY OUTCOMES:
margin-free (R0) resection rate | 1 years
  margin-free (R0) resection rate
3-year event-free survival rate | 3 years
  3-year event-free survival rate
safety, and quality of life | 1 year
  Adverse events (AEs) were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0.
3-year overall survival rate | 3 year
  3-year overall survival rate

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, MD, Principal Investigator — Cancer Center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cisel B, Pietrzak L, Michalski W, Wyrwicz L, Rutkowski A, Kosakowska E, Cencelewicz A, Spalek M, Polkowski W, Jankiewicz M, Stylinski R, Bebenek M, Kapturkiewicz B, Maciejczyk A, Sadowski J, Zygulska J, Zegarski W, Jankowski M, Las-Jankowska M, Toczko Z, Zelazowska-Omiotek U, Kepka L, Socha J, Wasilewska-Tesluk E, Markiewicz W, Kladny J, Majewski A, Kapuscinski W, Suwinski R, Bujko K; Polish Colorectal Study Group. Long-course preoperative chemoradiation versus 5 x 5 Gy and consolidation chemotherapy for clinical T4 and fixed clinical T3 rectal cancer: long-term results of the randomized Polish II study. Ann Oncol. 2019 Aug 1;30(8):1298-1303. doi: 10.1093/annonc/mdz186. PMID 31192355
- [Derived] Lin Z, Zhang P, Cai M, Li G, Liu T, Cai K, Wang J, Liu J, Liu H, Zhang W, Gao J, Wu C, Wang L, Wang Z, Hou Z, Kou H, Tao K, Zhang T. Neoadjuvant short-course radiotherapy followed by camrelizumab and chemotherapy for locally advanced rectal cancer: 3-year survival from a phase 2 study. BMC Med. 2025 May 9;23(1):273. doi: 10.1186/s12916-025-04087-x. PMID 40346524
- [Derived] Lin Z, Cai M, Zhang P, Li G, Liu T, Li X, Cai K, Nie X, Wang J, Liu J, Liu H, Zhang W, Gao J, Wu C, Wang L, Fan J, Zhang L, Wang Z, Hou Z, Ma C, Yang K, Wu G, Tao K, Zhang T. Phase II, single-arm trial of preoperative short-course radiotherapy followed by chemotherapy and camrelizumab in locally advanced rectal cancer. J Immunother Cancer. 2021 Nov;9(11):e003554. doi: 10.1136/jitc-2021-003554. PMID 34725214